CLINICAL TRIAL: NCT04051632
Title: Analysis of Glycemic Control in Type 1 Diabetes Patients Using Hybrid Closed Loop Insulin Pump Therapy (Medtronic 670G)
Status: Completed | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Gregory Goodwin, Senior Associate Physician in Medicine, Boston Children's Hospital
Other Study IDs: IRB-P00028472
Record Dates: First submitted 2019-08-06; First posted 2019-08-09 (Actual); Last update posted 2019-08-09 (Actual); Status verified 2019-08

CONDITIONS: Biomedical Technology; Type 1 Diabetes
Keywords: Medtronic 670G
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Type 1 Diabetes patients treated with the Medtronic 670G: Type 1 Diabetes patients treated with the Medtronic 670G at Boston Childrens Hospital
  Interventions: Device: Medtronic 670G insulin pump

INTERVENTIONS:
Device: Medtronic 670G insulin pump — * percent of patients who continue to use Medtronic 670G over time
  * impact of 670G on glycemic control: hemoglobin A1c, time in range

SUMMARY:
Observational study of patients at Boston Childrens Hospital with type 1 diabetes (T1D) who elected to treat their diabetes with the Medtronic 670 G hybrid closed loop insulin pump.

DETAILED DESCRIPTION:
Outcome study of 90-100 patients with type 1 diabetes who elected to use the Medtronic 670G.

Major outcome measure was to assess the percent of patients who were able to successfully continue to use the 670G technology over time.

Additional outcome variables included hemoglobin A1c pre and post treatment with the 670G, time in desired glucose range 70-180.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of T1D
* patient of Boston Childrens Hospital diabetes program
* deemed to be adequate candidates for hybrid closed loop technology by their diabetes health care team
* patient received Medtronic 670G training at Boston Childrens Hospital
* patient received follow up diabetes care at Boston Childrens Hospital for at least 3 months after starting on the 670G

Exclusion Criteria:

* patients not trained at Boston Childrens Hospital or self started

Ages: 5 Years to 25 Years | Sex: All
Age Groups: Child, Adult
Study Population: Single institution clinic population.
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2018-06-13 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
Successful implementation of hybrid closed loop technology | 0-24 months
  Percent of Type 1 Diabetes patients who were properly trained on the use of the 670G that continue to use Hybrid Closed Loop technology at 0, 6, 12, 18 and 24 months post training.

SECONDARY OUTCOMES:
Impact of hybrid closed loop technology on glycemic control | 0-24 months
  Assess impact of hybrid closed loop technology on glycemic control by comparing hemoglobin A1c measurements 0-6 months prior to treatment versus 0-6, 6-12, 12-18, 18-24 months post treatment
Assess impact of hybrid closed loop technology on glycemic control by analysis of sensor glucose data. | 0-24 months.
  Compare sensor glucose data: 1) percent time in range (70-180 mg/dl), 2)percent time in auto-mode, 3) percent time sensor usage versus hemoglobin A1c data over time.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Goodwin, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Childrens Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No